CLINICAL TRIAL: NCT07240415
Title: Extracorporeal Shockwave Therapy for Primary Lipedema: A Randomized Controlled Trial
Brief Title: ESWT for Primary Lipedema
Acronym: ESWT-LIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Bagcier (Other)
Responsible Party: Sponsor-Investigator, Fatih Bagcier, Associate Professor, Kars State Hospital
Organization: Kars State Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sba150585
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lipedema
Keywords: Lipedema; Extracorporeal Shockwave Therapy; ESWT; Radial Shockwave; Chronic Pain
MeSH Terms: conditions — Lipedema; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups receiving either standard conservative therapy alone or standard therapy plus radial ESWT. Outcome assessments will be performed by a blinded evaluator.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments, including VAS, SF-36, and circumference measurements, will be performed by an evaluator who is blinded to group allocation. Participants and treatment providers will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Conservative Therapy (Active Comparator): Participants receive standard conservative treatment including manual lymphatic drainage, pneumatic compression, Class II compression garments, and a home-based exercise program.
  Interventions: Other: Standard Conservative Therapy
- Standard Therapy plus ESWT (Experimental): Participants receive standard conservative treatment plus radial extracorporeal shockwave therapy (ESWT) applied twice weekly for 4 weeks (8 sessions) to the thighs and calves.
  Interventions: Other: Standard Conservative Therapy; Device: radial ESWT

INTERVENTIONS:
Other: Standard Conservative Therapy — Manual lymphatic drainage, pneumatic compression, Class II compression garments, and a home-based exercise program.
Device: radial ESWT — adial extracorporeal shockwave therapy using a BTL device (2.0-2.5 bar, 12 Hz, 1000 shocks per region, 20-mm head), twice weekly for 4 weeks (8 sessions).
  Arms: Standard Therapy plus ESWT

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of extracorporeal shockwave therapy (ESWT) when added to standard conservative treatment in women with primary lipedema. Participants will be randomly assigned to receive either standard conservative therapy alone or standard therapy combined with radial ESWT. The study will assess changes in pain intensity (VAS), limb circumference measurements, quality of life (SF-36), and patient satisfaction over an 8-week period. Evaluations will be performed at baseline, at the end of the 4-week treatment phase, and at 4-week follow-up. This trial seeks to provide evidence on whether ESWT offers additional clinical benefit in the management of primary lipedema.

DETAILED DESCRIPTION:
Lipedema is a chronic, progressive adipose tissue disorder characterized by disproportionate subcutaneous fat accumulation, pain, tenderness, easy bruising, and functional limitations. It predominantly affects women and leads to impaired mobility and reduced quality of life. Current international guidelines recommend conservative therapies as first-line management, including manual lymphatic drainage, pneumatic compression, compression garments, targeted exercise programs, and patient education. Although these interventions improve pain and function, their impact on underlying fibrotic changes and tissue stiffness is limited, creating a need for adjunctive treatments.

Extracorporeal shockwave therapy (ESWT) has been shown to enhance microcirculation, modulate inflammation, improve lymphatic flow, and exert anti-fibrotic effects through mechanotransduction. Positive outcomes have been reported in conditions with similar tissue characteristics, such as cellulite, lymphedema, and post-liposuction fibrosis. However, no randomized controlled trials have evaluated the efficacy of ESWT specifically in primary lipedema. This trial aims to address this gap in the literature.

This prospective, randomized, evaluator-blinded, controlled clinical study will include adult women aged 18-65 years diagnosed with Stage I-II primary lipedema according to Wold criteria. Eligible participants will be recruited from the Physical Medicine and Rehabilitation outpatient clinic of Medical Point Gaziantep Hospital. Participants will be randomized in a 1:1 ratio into two groups: (1) standard conservative therapy alone, or (2) standard conservative therapy plus radial ESWT. Conservative treatment will include manual lymphatic drainage, pneumatic compression therapy, Class II compression garments, and a home-based exercise program.

The ESWT group will receive additional radial ESWT using a BTL device with the following parameters: 2.0-2.5 bar pressure, 12 Hz frequency, 1000 shocks per region, 20-mm radial applicator head. Treatment regions will include the anterolateral thigh, medial thigh, and posterolateral calf. ESWT will be administered twice weekly for 4 weeks, totaling 8 sessions. Limb circumference will be measured at predefined anatomical points (thigh +10 cm/+20 cm above the patella, calf 10 cm above the medial malleolus, and ankle at the narrowest point).

Outcome measures will include pain intensity (VAS), quality of life (SF-36), limb circumference measurements, and patient satisfaction. Assessments will be performed at baseline (T0), immediately after completion of the 4-week intervention period (T1), and 4 weeks post-treatment (T2). The primary outcome is the change in VAS pain score from baseline to week 4. Secondary outcomes include changes in limb circumference, SF-36 scores, and satisfaction ratings, as well as the monitoring of any adverse events.

The study aims to determine whether adding ESWT to standard conservative management results in superior clinical outcomes compared with standard therapy alone. Findings may contribute to the development of evidence-based therapeutic strategies for women with primary lipedema.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18-65 years Diagnosis of primary lipedema (Stage I-II according to Wold criteria) Stable body weight for the past 3 months Ability to comply with compression garment use Willingness to participate and ability to provide informed consent

Exclusion Criteria:

Secondary lipedema or severe venous disease (CEAP C4 or higher) Liposuction or similar procedures within the past 6 months Pregnancy or breastfeeding Active infection, inflammation, or thrombosis Use of high-dose anticoagulants Contraindications to extracorporeal shockwave therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is limited to biological females because primary lipedema occurs almost exclusively in women.
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Limb Circumference Measurements | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Circumference will be measured at the thigh (+10 cm and +20 cm above the patella), calf (10 cm above the medial malleolus), and ankle (narrowest point). The change from baseline will be compared at Week 4 and Week 8.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst possible pain). The primary analysis will compare the change in VAS score between baseline and the end of the 4-week treatment period.
Short Form-36 Health Survey (SF-36) | Baseline (T0), Week 4 (T1), Week 8 (T2)
  Quality of life will be evaluated using the SF-36 questionnaire. Changes in physical and mental component scores will be assessed across time points.
Treatment Satisfaction (Likert Scale) | Week 4 (T1), Week 8 (T2)
  Patient satisfaction will be assessed using a 5-point Likert scale (1 = very dissatisfied to 5 = very satisfied).

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Result] Knobloch K, Kraemer R. Extracorporeal shock wave therapy (ESWT) for the treatment of cellulite--A current metaanalysis. Int J Surg. 2015 Dec;24(Pt B):210-7. doi: 10.1016/j.ijsu.2015.07.644. Epub 2015 Jul 22. PMID 26209782
- [Result] Knobloch K, Joest B, Kramer R, Vogt PM. Cellulite and focused extracorporeal shockwave therapy for non-invasive body contouring: a randomized trial. Dermatol Ther (Heidelb). 2013 Dec;3(2):143-55. doi: 10.1007/s13555-013-0039-5. Epub 2013 Dec 3. PMID 24297647
- [Result] Siems W, Grune T, Voss P, Brenke R. Anti-fibrosclerotic effects of shock wave therapy in lipedema and cellulite. Biofactors. 2005;24(1-4):275-82. doi: 10.1002/biof.5520240132. PMID 16403988